CLINICAL TRIAL: NCT05997290
Title: A PHASE 2/3 PROTOCOL TO INVESTIGATE THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF BNT162b2 RNA-BASED VACCINE CANDIDATES FOR SARS-CoV-2 NEW VARIANTS IN HEALTHY INDIVIDUALS
Brief Title: A Study to Learn About New COVD-19 RNA Vaccine Candidates for New Variants in Healthy Individuals
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: C4591054; 2024-000361-24 (Registry Identifier: EudraCT); NCT05997290 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2023-08-10; First posted 2023-08-18 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: SARS-CoV-2 Infection; COVID-19
Keywords: COVID-19; Coronavirus; Vaccine; SARS-CoV-2; RNA Vaccine; Vaccine-naïve
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — BNT162 Vaccine

STUDY DESIGN:
Intervention Model Description: Phase 2/3, controlled study
Masking Description: Open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- SSA: Group 1 (Experimental): Participants 12 years of age and older, COVID-19 vaccine-experienced will receive 30 µg of BNT162b2 (Omi XBB.1.5) at Visit 1.
  Interventions: Biological: BNT162b2 (Omi XBB.1.5)
- SSB: Group 2 (Experimental): Participants 12 years of age and older who were previously exposed to SARS-CoV-2 and are COVID-19 vaccine-naïve will receive 30 μg of BNT162b2 (Omi XBB.1.5) at Visit 1
  Interventions: Biological: BNT162b2 (Omi XBB.1.5)
- SSC: Group 3 (Experimental): Cohort 1 - Participants 18 years of age and older will receive 30 µg of BNT162b2 (Omi JN.1) at Visit 1.
  Interventions: Biological: BNT162b2 (Omi JN.1)
- SSC: Group 4 (Experimental): Cohort 2 - Participants 12 years of age and older will receive 30 µg of BNT162b2 (Omi JN.1) at Visit 1.
  Interventions: Biological: BNT162b2 (Omi JN.1)
- SSC - Group 5 (Experimental): Cohort 3 - Participants 18 years of age and older who will receive 30 µg of BNT162b2 (Omi KP.2) at Visit 1.
  Interventions: Biological: BNT162b2 (Omi KP.2)

INTERVENTIONS:
Biological: BNT162b2 (Omi XBB.1.5) — BNT162b2 monovalent (Omicron XBB.1.5)
  Arms: SSA: Group 1; SSB: Group 2
Biological: BNT162b2 (Omi JN.1) — BNT162b2 monovalent (Omicron JN.1)
  Arms: SSC: Group 3; SSC: Group 4
Biological: BNT162b2 (Omi KP.2) — BNT162b2 monovalent (Omicron KP.2)
  Arms: SSC - Group 5

SUMMARY:
The purpose of this clinical protocol is to learn about the safety, tolerability, and immunogenicity of new BNT162b2 RNA-based vaccine candidates targeting new variants of SARS-CoV-2 in healthy people.

Substudy A:

* This study will evaluate the safety, tolerability, and immunogenicity of BNT162b2 (Omi XBB.1.5) given as a single 30 µg dose,

  * in people who are 12 years of age and older,
  * who previously received at least 3 doses of a US-authorized mRNA COVID-19 vaccine, with the most recent dose being an Omicron BA.4/BA.5-adapted bivalent vaccine received at least 150 days before the study vaccination (Visit 1).
* The study is about 6 months long for each participant.
* Participants will have at least 5 visits to the clinic.
* At each clinic visit a blood sample will be taken.
* At least 1 nasal swab will taken.

Substudy B:

* This study will evaluate the safety, tolerability, and immunogenicity of BNT162b2 (Omi XBB.1.5) given as a single 30 µg dose,

  * in people who are 12 years of age and older,
  * who are COVID-19 vaccine-naïve
  * who have had any positive SARS-CoV-2 test result >28 days before study vaccine administration.
* The study is about 6 months long for each participant.
* Participants will have at least 5 visits to the clinic.
* At each clinic visit a blood sample will be taken.
* At least 1 nasal swab will taken.

Substudy C:

* This study will evaluate the safety, tolerability, and immunogenicity of BNT162b2 (Omi JN.1) and BNT162b2 (Omi KP.2) given as a single 30 µg dose to:

  * Cohort 1: people who are 18 years of age and older, who will receive BNT162b2 (Omi JN.1), and,
  * Cohort 2: people who are 12 years of age and older, who will receive BNT162b2 (Omi JN.1), and,
  * Cohort 3: people who are 18 years of age and older who will receive BNT162b2 (Omi KP.2).
  * Participants may have never received a COVID-19 vaccine or, may have previously received COVID-19 vaccine(s), with the most recent dose received at least 150 days before the study vaccination (Visit 1).
* The study is about 6 months long for each participant.
* Participants will have at least 6 visits (Cohorts 1 and 3) or at least 5 visits (Cohort 2) to the clinic.
* At each clinic visit a blood sample will be taken.
* At least 1 nasal swab will taken.

ELIGIBILITY:
SSA

Inclusion Criteria:

* Received at least 3 prior doses of a US-authorized mRNA COVID-19 vaccine, with the most recent dose being a US-authorized Omicron BA.4/BA.5-adapted bivalent vaccine received at least 150 days before Visit 1 (Day 1).
* 12 years of age and older
* Healthy participants (stable pre-existing disease permitted).
* Willing and able to comply with all scheduled visits/contacts, study procedures and lifestyle considerations.
* Capable of giving, or parent(s)/legal guardian capable of giving, signed informed consent.

Exclusion Criteria

* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study vaccines.
* Immunocompromised with known or suspected immunodeficiency, as determined by history and/or laboratory/physical examination.
* Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.
* Women who are pregnant or breastfeeding.
* Any medical or psychiatric condition, or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* History of myocarditis or pericarditis.
* Receipt of systemic treatment with known immunosuppressant medications (including cytotoxic agents or systemic corticosteroids, eg, for cancer or an autoimmune disease), or radiotherapy, within 60 days before enrollment or planned receipt through conclusion of the study.
* Receipt of blood/plasma products, immunoglobulin, or monoclonal antibodies, used for the treatment or prevention of COVID-19 or those that are considered immunosuppressive, from 60 days before study vaccination or planned receipt throughout the study.
* Participation in other studies involving receipt of other study intervention within 28 days before enrollment. Anticipated participation in other studies involving other study intervention from enrollment through the end of this study.
* Investigator site staff directly involved in the conduct of the study and their family members, site staff otherwise supervised by the investigator, and sponsor and sponsor delegate employees directly involved in the conduct of the study and their family members.

SSB

Inclusion Criteria:

* COVID-19 vaccine-naïve.
* Any positive SARS-CoV-2 test result >28 days before study intervention administration.
* 12 years of age and older.
* Healthy participants (stable pre-existing disease permitted).
* Willing and able to comply with all scheduled visits/contacts, study procedures and lifestyle considerations.
* Capable of giving or parent(s)/legal guardian capable of giving, signed informed consent.

Exclusion Criteria:

* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study vaccines.
* Immunocompromised individuals with known or suspected immunodeficiency, as determined by history and/or laboratory/physical examination.
* Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.
* Women who are pregnant or breastfeeding.
* Any medical or psychiatric condition, including recent (within the past year) or active suicidal ideation/behavior, or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* History of myocarditis or pericarditis.
* Receipt of systemic treatment with known immunosuppressant medications (including cytotoxic agents or systemic corticosteroids*, eg, for cancer or an autoimmune disease), or radiotherapy, within 60 days before enrollment or planned receipt through conclusion of the study.
* Receipt of blood/plasma products, immunoglobulin, or monoclonal antibodies used for the treatment or prevention of COVID-19 or those that are considered immunosuppressive, from 60 days before study intervention administration or planned receipt throughout the study.
* Participation in other studies involving receipt of other study intervention within 28 days before enrollment. Anticipated participation in other studies involving other study intervention from enrollment through the end of this study.
* Investigator site staff directly involved in the conduct of the study and their family members, site staff otherwise supervised by the investigator, and sponsor and sponsor delegate employees directly involved in the conduct of the study and their family members.

SSC

Inclusion Criteria:

* Cohort 1: 18 years of age and older
* Cohort 2: 12 years of age and older
* Cohort 3: 18 years of age and older
* Healthy participants (stable pre-existing disease permitted).
* Willing and able to comply with all scheduled visits/contacts, study procedures and lifestyle considerations.
* Capable of giving, or parent(s)/legal guardian capable of giving, signed informed consent.

Exclusion Criteria

* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study vaccines.
* Immunocompromised with known or suspected immunodeficiency, as determined by history and/or laboratory/physical examination.
* Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.
* Women who are pregnant or breastfeeding.
* Any medical or psychiatric condition, or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* History of myocarditis or pericarditis.
* Receipt of systemic treatment with known immunosuppressant medications (including cytotoxic agents or systemic corticosteroids, eg, for cancer or an autoimmune disease), or radiotherapy, within 60 days before enrollment or planned receipt through conclusion of the study.
* Receipt of blood/plasma products, immunoglobulin, or monoclonal antibodies, used for the treatment or prevention of COVID-19 or those that are considered immunosuppressive, from 60 days before study vaccination or planned receipt throughout the study.
* Receipt of a COVID-19 vaccine less than 150 days before study intervention administration Visit 1 (Day 1).
* Participation in other studies involving receipt of other study intervention within 28 days before enrollment. Anticipated participation in other studies involving other study intervention from enrollment through the end of this study.
* Investigator site staff directly involved in the conduct of the study and their family members, site staff otherwise supervised by the investigator, and sponsor and sponsor delegate employees directly involved in the conduct of the study and their family members.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1051 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2025-03-13 (Actual); Study Completion 2025-03-13 (Actual)

PRIMARY OUTCOMES:
SSA: Percentage of participants reporting local reactions | For up to 7 days following the study vaccination
  Pain at the injection site, redness, and swelling, as self-reported in electronic diaries.
SSA: Percentage of participants reporting systemic events | For up to 7 days following the study vaccination
  Fever, fatigue, headache, chills, vomiting, diarrhea, new or worsened muscle pain, and new or worsened joint pain, as self-reported in electronic diaries
SSA: Percentage of participants reporting adverse events | Through 1 month after the study vaccination
  As elicited by the investigational staff
SSA: Percentage of participants reporting serious adverse events | Through 6 months after the study vaccination
  As elicited by the investigational staff
SSA: Geometric Mean Titers (GMT) of SARS-CoV-2 Omicron XBB.1.5- and Omicron BA.4/BA.5-neutralizing antibody levels for BNT162b2 (Omi XBB.1.5) 30 µg | At 1 month after the study vaccination
  As measured at the central laboratory
SSA: Geometric Mean Fold Rise (GMFR; change between 2 timepoints) of SARS-CoV-2 Omicron XBB.1.5-and Omicron BA.4/BA.5-neutralizing antibody levels for BNT162b2 (Omi XBB.1.5) 30 µg | From before study vaccination (Day 1) to 1 month after study vaccination
  As measured at the central laboratory
SSA: Percentages of participants with seroresponse to BNT162b2 (Omi XBB.1.5) 30 µg in terms of GMTs of SARS-CoV-2 Omicron XBB.1.5- and Omicron BA.4/BA.5-neutralizing antibody levels | At 1 month after the study vaccination
  As measured at the central laboratory
SSB: Percentage of participants reporting local reactions | For up to 7 days following the study vaccination
  Pain at the injection site, redness, and swelling, as self-reported in electronic diaries.
SSB: Percentage of participants reporting systemic events | For up to 7 days following the study vaccination
  Fever, fatigue, headache, chills, vomiting, diarrhea, new or worsened muscle pain, and new or worsened joint pain, as self-reported in electronic diaries.
SSB: Percentage of participants reporting adverse events | Through 1 month after the study vaccination
  As elicited by the investigational staff.
SSB: Percentage of participants reporting serious adverse events | Through 6 months after the study vaccination
  As elicited by the investigational staff.
SSB: Geometric Mean Ratio (GMR) of the SARS-CoV-2 XBB.1.5-neutralizing titers after BNT162b2 (Omi XBB.1.5) 30 μg given as single dose to COVID-19 vaccine-naïve subjects to BNT162b2 (Omi XBB.1.5) 30 μg given to vaccine-experienced participants in SSA. | At 1 month after vaccination.
  As measured at the central laboratory
Difference in percentages of subjects with seroresponse to XBB.1.5 strain after BNT162b2 (Omi XBB.1.5) 30 μg given as single dose to COVID-19 vaccine-naïve subjects compared to BNT162b2 (Omi XBB.1.5) 30 μg given to vaccine experienced subjects in SSA | At 1 month after vaccination
  As measured at the central laboratory
SSC Cohort 1 and Cohort 2 combined: Percentage of participants reporting local reactions | For up to 7 days following the study vaccination
  Pain at the injection site, redness, and swelling, as self-reported in electronic diaries.
SSC Cohort 1 and Cohort 2 combined: Percentage of participants reporting systemic events | For up to 7 days following the study vaccination
  Fever, fatigue, headache, chills, vomiting, diarrhea, new or worsened muscle pain, and new or worsened joint pain, as self-reported in electronic diaries
SSC Cohort 1 and Cohort 2 combined: Percentage of participants reporting adverse events | Through 1 month after the study vaccination
  As elicited by the investigational staff
SSC Cohort 1 and Cohort 2 combined: Percentage of participants reporting serious adverse events | Through 6 months after the study vaccination
  As elicited by the investigational staff
SSC Cohort 1 and Cohort 2 combined: Geometric Mean Titers (GMT) of SARS-CoV-2 Omicron JN.1- and Omicron XBB.1.5- neutralizing antibody levels for BNT162b2 (Omi JN.1) 30 µg. | At 1 month after the study vaccination
  As measured at the central laboratory
SSC Cohort 1 and Cohort 2 combined: Geometric Mean Fold Rise (GMFR; change between 2 timepoints) of SARS-CoV-2 Omicron JN.1- and Omicron XBB.1.5- neutralizing antibody levels for BNT162b2 (Omi JN.1) 30 µg. | From before study vaccination (Day 1) to 1 month after study vaccination
  As measured at the central laboratory
SSC Cohort 1 and Cohort 2 combined: Percentages of participants with seroresponse to BNT162b2 (Omi JN.1) 30 µg in terms of GMTs of SARS-CoV-2 Omicron JN.1- and Omicron XBB.1.5-neutralizing antibody levels. | At 1 month after the study vaccination
  As measured at the central laboratory
SSC Cohort 3: Percentage of participants reporting local reactions | For up to 7 days following the study vaccination
  Pain at the injection site, redness, and swelling, as self-reported in electronic diaries.
SSC Cohort 3: Percentage of participants reporting systemic events | For up to 7 days following the study vaccination
  Fever, fatigue, headache, chills, vomiting, diarrhea, new or worsened muscle pain, and new or worsened joint pain, as self-reported in electronic diaries
SSC Cohort 3: Percentage of participants reporting adverse events | Through 1 month after the study vaccination
  As elicited by the investigational staff
SSC Cohort 3: Percentage of participants reporting serious adverse events | Through 6 months after the study vaccination
  As elicited by the investigational staff
SSC Cohort 3: Geometric Mean Titers (GMT) of SARS-CoV-2 Omicron KP.2- and Omicron JN.1- neutralizing antibody levels for BNT162b2 (Omi KP.2) 30 µg. | At 1 month after the study vaccination
  As measured at the central laboratory
SSC Cohort 3: Geometric Mean Fold Rise (GMFR; change between 2 timepoints) of SARS-CoV-2 Omicron KP.2- and Omicron JN.1- neutralizing antibody levels for BNT162b2 (Omi KP.2) 30 µg. | From before study vaccination (Day 1) to 1 month after study vaccination
  As measured at the central laboratory
SSC Cohort 3: Percentages of participants with seroresponse to BNT162b2 (Omi KP.2) 30 µg in terms of GMTs of SARS-CoV-2 Omicron KP.2- and Omicron JN.1- neutralizing antibody levels. | At 1 month after the study vaccination
  As measured at the central laboratory

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (36):
- United States (36):
  - North Alabama Research Center, Athens, Alabama
  - Medical Affiliated Research Center, Huntsville, Alabama
  - Alliance for Multispecialty Research, LLC, Mobile, Alabama
  - Epic Medical Research - Surprise, Surprise, Arizona
  - Alliance for Multispecialty Research, LLC, Tempe, Arizona
  - West Coast Research, Dublin, California
  - California Research Foundation, San Diego, California
  - Bayview Research Group, LLC, Valley Village, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Clinical Research Consulting, Milford, Connecticut
  - Indago Research & Health Center, Inc, Hialeah, Florida
  - Clinical Neuroscience Solutions, Inc. dba CNS Healthcare, Jacksonville, Florida
  - Care Research - West Flagler Street, Miami, Florida
  - Acevedo Clinical Research Associates, Miami, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Clinical Research Atlanta, Stockbridge, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Kentucky Pediatric/ Adult Research, Bardstown, Kentucky
  - Bio-Kinetic Clinical Applications, LLC dba QPS-MO, Springfield, Missouri
  - Bio-Kinetic Clinical Applications LLC DBA QPS_MO (Patient Screening Only), Springfield, Missouri
  - M3 Wake Research, Inc., Raleigh, North Carolina
  - Centricity Research Columbus Ohio Multispecialty, Columbus, Ohio
  - Dayton Clinical Research, Dayton, Ohio
  - Senders Pediatrics, South Euclid, Ohio
  - Alliance for Multispecialty Research, LLC, Knoxville, Tennessee
  - Clinical Neuroscience Solutions Inc., Memphis, Tennessee
  - Zenos Clinical Research, Dallas, Texas
  - Epic Medical Research - DeSoto, DeSoto, Texas
  - DM Clinical Research - Bellaire, Houston, Texas
  - SMS Clinical Research, Mesquite, Texas
  - IMA Clinical Research San Antonio, San Antonio, Texas
  - DM Clinical Research, Tomball, Texas
  - Alliance for Multispecialty Research, LLC, Layton, Utah
  - J. Lewis Research, Inc. / Foothill Family Clinic, Salt Lake City, Utah
  - J. Lewis Research, Inc. / Foothill Family Clinic South, Salt Lake City, Utah
  - Alliance for Multispecialty Research, LLC, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Diya O, Gayed J, Lowry FS, Ma H, Bangad V, Mensa F, Zou J, Xie X, Hu Y, Cutler M, Belanger T, Cooper D, Xu X, Mogg R, Tureci O, Sahin U, Swanson KA, Modjarrad K, Anderson AS, Gurtman A, Kitchin N. Safety and Immunogenicity of Monovalent Omicron KP.2-Adapted BNT162b2 COVID-19 Vaccine in Adults: Single-Arm Substudy from a Phase 2/3 Trial. Infect Dis Ther. 2025 Aug;14(8):1973-1987. doi: 10.1007/s40121-025-01185-4. Epub 2025 Jul 1. PMID 40591130
- [Derived] Diya O, Gayed J, Lowry FS, Ma H, Bangad V, Mensa F, Zou J, Xie X, Hu Y, Cutler M, Belanger T, Cooper D, Xu X, Koury K, Tureci O, Sahin U, Swanson KA, Modjarrad K, Anderson AS, Gurtman A, Kitchin N. A phase 2/3 trial to investigate the safety and immunogenicity of monovalent Omicron JN.1-adapted BNT162b2 COVID-19 vaccine in adults >/=18 years old. Vaccine. 2025 Apr 11;52:126869. doi: 10.1016/j.vaccine.2025.126869. Epub 2025 Feb 24. PMID 39999538
- [Derived] Gayed J, Bangad V, Xu X, Mensa F, Cutler M, Tureci O, Sahin U, Modjarrad K, Swanson KA, Anderson AS, Gurtman A, Kitchin N; C4591054 Study Group. Immunogenicity of the Monovalent Omicron XBB.1.5-Adapted BNT162b2 COVID-19 Vaccine against XBB.1.5, BA.2.86, and JN.1 Sublineages: A Phase 2/3 Trial. Vaccines (Basel). 2024 Jul 2;12(7):734. doi: 10.3390/vaccines12070734. PMID 39066372
- [Derived] Gayed J, Diya O, Lowry FS, Xu X, Bangad V, Mensa F, Zou J, Xie X, Hu Y, Lu C, Cutler M, Belanger T, Cooper D, Koury K, Anderson AS, Tureci O, Sahin U, Swanson KA, Modjarrad K, Gurtman A, Kitchin N; C4591054 Study Group. Safety and Immunogenicity of the Monovalent Omicron XBB.1.5-Adapted BNT162b2 COVID-19 Vaccine in Individuals >/=12 Years Old: A Phase 2/3 Trial. Vaccines (Basel). 2024 Jan 24;12(2):118. doi: 10.3390/vaccines12020118. PMID 38400102
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4591054